CLINICAL TRIAL: NCT06414759
Title: Efficacy and Safety of Combination Diuretic Therapy in Patients With Acute Decompensated Heart Failure and Volume Overload
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Ahmed Naguib Mohamed Abdelmoaty, Teaching Assistant of Clinical Pharmacy, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL3575; IHC00077 (Registry Identifier: General Organization for Teaching Hospitals and Institutes (GOTHI))
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Acute Decompensated Heart Failure; Volume Overload; Edema
Keywords: ADHF; Acute Decompensated Heart Failure; AHF; Acute Heart Failure; Volume overload; Edema; Loop diuretics; Fusrosemide; Metolazone; Acetazolamide; Carbonic anhydrase inhibitor; Thiazide like diuretics; Thiazide diuretics
MeSH Terms: conditions — Edema | interventions — Acetazolamide; Carbonic Anhydrase Inhibitors; Metolazone; Thiazides; Sodium Potassium Chloride Symporter Inhibitors

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-blinded, controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): First group (IV loop Diuretics + oral acetazolamide): patients will receive IV loop diuretic 2 times the outpatient oral (PO) daily dose, and oral loop diuretics will be stopped. In cases where the patient was not previously on oral diuretics, a starting dose of 40 mg of IV furosemide, IV bumetanide 1 mg or a bolus of 20 mg of IV torsemide can be utilized, together with acetazolamide: 500 mg PO once daily.
  Interventions: Drug: Acetazolamide; Drug: IV Loop Diuretics
- Group 2 (Experimental): Second group (IV loop diuretics + oral metolazone): patients will receive IV loop diuretic approximately 2 times the outpatient oral daily dose, and oral loop diuretics will be stopped. In cases where the patient was not previously on oral diuretics, a starting dose of 40 mg of IV furosemide, IV bumetanide 1 mg or a bolus of 20 mg of IV torsemide can be utilized, together with metolazone: 5 mg PO once daily.
  Interventions: Drug: Metolazone; Drug: IV Loop Diuretics

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide is a medication that belongs to the class of carbonic anhydrase inhibitors. It acts by reducing the reabsorption of sodium in the proximal tubules of the kidneys. When combined with loop diuretics, acetazolamide has the potential to enhance the effectiveness of diuretic therapy, thus aiding in the process of decongestion.
  It will be given 500mg orally, once daily.
  Other Names: Carbonic anhydrase inhibitor
  Arms: Group 1
Drug: Metolazone — Metolazone is a medication with properties like thiazide diuretics, prescribed for the management of congestive heart failure and hypertension. Its mechanism of action involves blocking the transport of sodium across the epithelium of renal tubules, predominantly in the distal tubules.
  It will be given 5mg orally, once daily.
  Other Names: Thiazide like diuretic
  Arms: Group 2
Drug: IV Loop Diuretics — IV loop diuretic 2 times the outpatient oral (PO) daily dose, and oral loop diuretics will be stopped. In cases where the patient was not previously on oral diuretics, a starting dose of 40 mg of IV furosemide, IV bumetanide 1 mg or a bolus of 20 mg of IV torsemide can be utilized.

SUMMARY:
This study aims to compare two medications, acetazolamide and metolazone, along with loop diuretics, to see which one works better and is safer for patients with ADHF who have volume overload. By comparing these medications, we hope to learn which one can help these patients the most. This will help doctors choose the best treatment for patients with ADHF and volume overload.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with ages ≥ 18 years old, and less than 65 years old.
* For both elective and emergency hospital admissions, patients with a clinical diagnosis of ADHF must exhibit at least one clinical sign indicative of volume overload. These signs may include edema (score 2 or higher), ascites confirmed through echography, or pleural effusion confirmed by chest X-ray or echography or rales on auscultation, or jugular venous pressure greater than10 mm Hg.

Exclusion Criteria:

* Patient diagnosed with acute kidney injury upon hospital admission based on the presence of any of the following criteria: an increase in SCr by at least 0.3 mg/dL within 48 hours, an increase in SCr to at least 2 times the baseline value, known or presumed to have occurred within the prior 7 days, and a urine volume less than 0.5 ml/kg/hour for a duration of 6 hours.
* Patients with acute pulmonary edema caused by increased afterload and fluid redistribution to the lungs in the absence or with minimal fluid accumulation.
* Anticipated exposure to nephrotoxic agents (such as contrast dye) during hospitalization.
* Patients who exhibit anuria or are undergoing renal replacement therapy or ultrafiltration.
* Patients with eGFR less than 30 mL/min/1.73m² at the time of screening.
* Expected use of intravenous inotropes, vasopressors, or nitroprusside during the study.
* Prior cardiac transplantation and/or utilization of a ventricular assist device.
* Blood pressure below 90 mmHg or mean arterial pressure below 65 mmHg at the time of recruitment.
* Patients who are pregnant or breastfeeding.
* Administration of acetazolamide or metolazone within the one-month period preceding randomization.
* The usage of any diuretic agent during the treatment phase is not specified in the study protocol, except for mineralocorticoid receptor antagonists.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Urine Output | 48 Hours
  Total Urine output Volume

SECONDARY OUTCOMES:
Diuretic Response | 48 Hours
  Urine output/40 mg furosemide equivalent
Body Weight | 48 Hours
  Change in Body Weight
Congestion Score | 48 Hours
  Change in congestion score (Modified ADVOR Trial Congestion Score)
NT-proBNP/BNP | On admission and before discharge (After 48 hours)
  Change in NT-Pro BNP/BNP levels
Bicarbonate Level | 48 Hours
  Change in bicarbonate level from baseline [VBG]
Serum Creatinine | 48 Hours
  Change in serum creatinine (SCr)
eGFR | 48 Hours
  Change in estimated glomerular filtration rate (eGFR) from baseline
Blood Pressure | 48 Hours
  Change in systolic blood pressure (SBP) from baseline
Potassium Level | 48 Hours
  Change in potassium level from baseline [VBG]
Length of Hospital Stay | Up to 2 weeks
  Both general ward and CCU
Mortality or HF Events | 3 Months
  All-cause mortality and heart failure readmission during 3 months of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Institute, Giza, GZ, Egypt

REFERENCES:
- [Background] Arrigo M, Jessup M, Mullens W, Reza N, Shah AM, Sliwa K, Mebazaa A. Acute heart failure. Nat Rev Dis Primers. 2020 Mar 5;6(1):16. doi: 10.1038/s41572-020-0151-7. PMID 32139695
- [Background] Njoroge JN, Teerlink JR. Pathophysiology and Therapeutic Approaches to Acute Decompensated Heart Failure. Circ Res. 2021 May 14;128(10):1468-1486. doi: 10.1161/CIRCRESAHA.121.318186. Epub 2021 May 13. PMID 33983837
- [Background] Hsiao R, Greenberg B. Contemporary Treatment of Acute Heart Failure. Prog Cardiovasc Dis. 2016 Jan-Feb;58(4):367-78. doi: 10.1016/j.pcad.2015.12.005. Epub 2016 Jan 5. PMID 26764279
- [Background] Kurmani S, Squire I. Acute Heart Failure: Definition, Classification and Epidemiology. Curr Heart Fail Rep. 2017 Oct;14(5):385-392. doi: 10.1007/s11897-017-0351-y. PMID 28785969
- [Background] Rubio-Gracia J, Demissei BG, Ter Maaten JM, Cleland JG, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, Davison BA, Givertz MM, Bloomfield DM, Dittrich H, Damman K, Perez-Calvo JI, Voors AA. Prevalence, predictors and clinical outcome of residual congestion in acute decompensated heart failure. Int J Cardiol. 2018 May 1;258:185-191. doi: 10.1016/j.ijcard.2018.01.067. PMID 29544928
- [Background] Mentz RJ, Kjeldsen K, Rossi GP, Voors AA, Cleland JG, Anker SD, Gheorghiade M, Fiuzat M, Rossignol P, Zannad F, Pitt B, O'Connor C, Felker GM. Decongestion in acute heart failure. Eur J Heart Fail. 2014 May;16(5):471-82. doi: 10.1002/ejhf.74. Epub 2014 Mar 5. PMID 24599738
- [Background] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Background] Hoorn EJ, Ellison DH. Diuretic Resistance. Am J Kidney Dis. 2017 Jan;69(1):136-142. doi: 10.1053/j.ajkd.2016.08.027. Epub 2016 Nov 1. PMID 27814935
- [Background] Suri SS, Pamboukian SV. Optimal diuretic strategies in heart failure. Ann Transl Med. 2021 Mar;9(6):517. doi: 10.21037/atm-20-4600. PMID 33850914
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Sica DA. Metolazone and its role in edema management. Congest Heart Fail. 2003 Mar-Apr;9(2):100-5. doi: 10.1111/j.1527-5299.2003.01907.x. PMID 12671341
- [Background] Cox ZL, Hung R, Lenihan DJ, Testani JM. Diuretic Strategies for Loop Diuretic Resistance in Acute Heart Failure: The 3T Trial. JACC Heart Fail. 2020 Mar;8(3):157-168. doi: 10.1016/j.jchf.2019.09.012. Epub 2019 Dec 11. PMID 31838029
- [Background] Verbrugge FH, Dupont M, Bertrand PB, Nijst P, Penders J, Dens J, Verhaert D, Vandervoort P, Tang WH, Mullens W. Determinants and impact of the natriuretic response to diuretic therapy in heart failure with reduced ejection fraction and volume overload. Acta Cardiol. 2015 Jun;70(3):265-73. doi: 10.1080/ac.70.3.3080630. PMID 26226699
- [Background] Verbrugge FH, Martens P, Ameloot K, Haemels V, Penders J, Dupont M, Tang WHW, Droogne W, Mullens W. Acetazolamide to increase natriuresis in congestive heart failure at high risk for diuretic resistance. Eur J Heart Fail. 2019 Nov;21(11):1415-1422. doi: 10.1002/ejhf.1478. Epub 2019 May 9. PMID 31074184
- [Background] Mullens W, Dauw J, Martens P, Verbrugge FH, Nijst P, Meekers E, Tartaglia K, Chenot F, Moubayed S, Dierckx R, Blouard P, Troisfontaines P, Derthoo D, Smolders W, Bruckers L, Droogne W, Ter Maaten JM, Damman K, Lassus J, Mebazaa A, Filippatos G, Ruschitzka F, Dupont M; ADVOR Study Group. Acetazolamide in Acute Decompensated Heart Failure with Volume Overload. N Engl J Med. 2022 Sep 29;387(13):1185-1195. doi: 10.1056/NEJMoa2203094. Epub 2022 Aug 27. PMID 36027559
- [Background] Mullens W, Damman K, Harjola VP, Mebazaa A, Brunner-La Rocca HP, Martens P, Testani JM, Tang WHW, Orso F, Rossignol P, Metra M, Filippatos G, Seferovic PM, Ruschitzka F, Coats AJ. The use of diuretics in heart failure with congestion - a position statement from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2019 Feb;21(2):137-155. doi: 10.1002/ejhf.1369. Epub 2019 Jan 1. PMID 30600580
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Jung B, Martinez M, Claessens YE, Darmon M, Klouche K, Lautrette A, Levraut J, Maury E, Oberlin M, Terzi N, Viglino D, Yordanov Y, Claret PG, Bige N; Societe de Reanimation de Langue Francaise (SRLF); Societe Francaise de Medecine d'Urgence (SFMU). Diagnosis and management of metabolic acidosis: guidelines from a French expert panel. Ann Intensive Care. 2019 Aug 15;9(1):92. doi: 10.1186/s13613-019-0563-2. PMID 31418093
- [Background] Kim HN, Januzzi JL Jr. Natriuretic peptide testing in heart failure. Circulation. 2011 May 10;123(18):2015-9. doi: 10.1161/CIRCULATIONAHA.110.979500. No abstract available. PMID 21555724
- [Background] Januzzi JL, van Kimmenade R, Lainchbury J, Bayes-Genis A, Ordonez-Llanos J, Santalo-Bel M, Pinto YM, Richards M. NT-proBNP testing for diagnosis and short-term prognosis in acute destabilized heart failure: an international pooled analysis of 1256 patients: the International Collaborative of NT-proBNP Study. Eur Heart J. 2006 Feb;27(3):330-7. doi: 10.1093/eurheartj/ehi631. Epub 2005 Nov 17. PMID 16293638
- [Background] Inker LA, Eneanya ND, Coresh J, Tighiouart H, Wang D, Sang Y, Crews DC, Doria A, Estrella MM, Froissart M, Grams ME, Greene T, Grubb A, Gudnason V, Gutierrez OM, Kalil R, Karger AB, Mauer M, Navis G, Nelson RG, Poggio ED, Rodby R, Rossing P, Rule AD, Selvin E, Seegmiller JC, Shlipak MG, Torres VE, Yang W, Ballew SH, Couture SJ, Powe NR, Levey AS; Chronic Kidney Disease Epidemiology Collaboration. New Creatinine- and Cystatin C-Based Equations to Estimate GFR without Race. N Engl J Med. 2021 Nov 4;385(19):1737-1749. doi: 10.1056/NEJMoa2102953. Epub 2021 Sep 23. PMID 34554658
- [Background] Ng TM, Konopka E, Hyderi AF, Hshieh S, Tsuji Y, Kim BJ, Han SY, Phan DH, Jeng AI, Lou M, Elkayam U. Comparison of bumetanide- and metolazone-based diuretic regimens to furosemide in acute heart failure. J Cardiovasc Pharmacol Ther. 2013 Jul;18(4):345-53. doi: 10.1177/1074248413482755. Epub 2013 Mar 27. PMID 23538300